CLINICAL TRIAL: NCT03784859
Title: Tissue Expansion in Breast Reconstruction Without Drains: A Study Using a Tissue Expander That Collects Periprosthetic Fluid
Brief Title: Tissue Expansion in Breast Reconstruction Without Drains
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Tiger Biosciences, LLC. (Industry)
Responsible Party: Principal Investigator, Edward Ray, Staff Physician II, Cedars-Sinai Medical Center
Other Study IDs: Pro00052823
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Hereditary Breast and Ovarian Cancer Syndrome; Breast Implant; Complications
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All patients in study: 5 consecutive patients with breast cancer or a breast cancer-causing gene that elect to undergo bilateral breast reconstruction will be Insertion of Tissue Expander with Fluid Reservoir as the first stage of reconstruction. Post-surgical care will be similar as patients with conventional expanders, except that during office visits, fluid will be transcutaneously aspirated from the fluid reservoir on each side.
  Interventions: Device: Insertion of Tissue Expander with Fluid Reservoir

INTERVENTIONS:
Device: Insertion of Tissue Expander with Fluid Reservoir — Use of unique expander type in first stage of a two-stage breast reconstruction, without prolonged drain placement.
  Other Names: Sientra AlloX2 Expander

SUMMARY:
The primary objective of this small feasibility pilot study is to demonstrate that implant-based breast reconstruction (after treatment for cancer) can successfully be performed without prolonged drain placement, using a tissue expander with a reservoir and in-office transcutaneous fluid aspiration. Secondly, the investigators aim to provide enough confidence in this technique that a larger study can be performed to demonstrate fewer complications (infection, drain-related pain and re-operation rates) when compared to the use of conventional tissue expanders and/or implants with prolonged drain placement.

DETAILED DESCRIPTION:
Patients electing to have staged, implant-based, bilateral breast reconstruction at the time of mastectomy (for either cancer or cancer prevention) will undergo a standardized subpectoral tissue expander placement (using the Sientra AlloX2 dual-port device) on each side of the chest with a single piece of acellular dermal matrix (ADM). A single drain in the subcutaneous pocket of each breast will be used and removed on the first post-operative day. Patients will be admitted for overnight observation in the hospital. Each post-operative day fluid will be aspirated from each reservoir port using a standard sterile technique, and the volume recorded. After discharge, patients will be seen in the office within one week of discharge and fluid aspirated from each expander using the reservoir ports, and the volume shall be recorded. The aspiration will be repeated weekly until expansion is completed and/or the amount of fluid aspirated is less than 10 cc.

Patients will be asked to complete a 7 item multiple-choice questionnaire regarding their attitudes about their breast reconstruction, first at completion of tissue expansion and finally at their first follow-up visit following placement of permanent breast implants.

This study utilizes FDA 510k-classified devices that allow removal of fluid without drains, in lieu of more conventional expanders, allowing for the avoidance of prolonged drain usage.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bilateral breast reconstruction following mastectomy (performed to treat stage I-III breast cancer or for prevention of breast cancer).
* Non-smokers
* BMI less than 31
* No other significant surgical risk factors that make elective use of implants dangerous (e.g., presence of a pacemaker, frail health, dependence on blood thinners, uncontrolled diabetes, bleeding tendencies, autoimmune disorders, immune compromise)

Exclusion Criteria:

* Unilateral mastectomy patients
* Current smokers
* Those with bleeding dyscrasias or clotting disorders
* Those who have had or will have a full axillary lymph node dissection
* Cases where there is an unusually high degree of bleeding intra-operatively (more than 150 cc)
* Those with a BMI greater than 30
* Those with history of prior breast surgery (aside from lumpectomy or needle biopsy)
* Those with a history of prior breast radiation
* Those with stage IV or unresectable breast cancer
* Significant surgical risk factors that make elective use of implants dangerous (e.g., presence of a pacemaker, frail health, dependence on blood thinners, uncontrolled diabetes, bleeding tendencies, autoimmune disorders, immune compromise)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients are usually candidates for reconstruction using breast implants
Study Population: Women over the age of 21 with breast cancer or a gene that increases the risk of breast cancer who elect to undergo bilateral mastectomies and two-stage implant-based reconstruction using tissue expanders and permanent implants.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with successful breast reconstruction using reservoir-expanders | 4-6 months
  The number of patients that successfully complete two stage implant-based breast reconstruction with fluid-reservoir tissue expanders and early drain removal. An outcome failure would be if the expander required removal due to uncontrolled seroma, infection or other factor that prevents a successful implant-based reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Ray, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith JM, Broyles JM, Guo Y, Tuffaha SH, Mathes D, Sacks JM. Human acellular dermis increases surgical site infection and overall complication profile when compared with submuscular breast reconstruction: An updated meta-analysis incorporating new products✰. J Plast Reconstr Aesthet Surg. 2018 Nov;71(11):1547-1556. doi: 10.1016/j.bjps.2018.06.012. Epub 2018 Jul 6. PMID 30093286
- [Background] Kim JYS, Davila AA, Persing S, Connor CM, Jovanovic B, Khan SA, Fine N, Rawlani V. A meta-analysis of human acellular dermis and submuscular tissue expander breast reconstruction. Plast Reconstr Surg. 2012 Jan;129(1):28-41. doi: 10.1097/PRS.0b013e3182361fd6. PMID 22186498
- [Background] Ollech CJ, Block LM, Afifi AM, Poore SO. Effect of Drain Placement on Infection, Seroma, and Return to Operating Room in Expander-Based Breast Reconstruction. Ann Plast Surg. 2017 Dec;79(6):536-540. doi: 10.1097/SAP.0000000000001174. PMID 28671886
- [Background] Srivastava V, Basu S, Shukla VK. Seroma formation after breast cancer surgery: what we have learned in the last two decades. J Breast Cancer. 2012 Dec;15(4):373-80. doi: 10.4048/jbc.2012.15.4.373. Epub 2012 Dec 31. PMID 23346164
- [Background] Sampathraju S, Rodrigues G. Seroma formation after mastectomy: pathogenesis and prevention. Indian J Surg Oncol. 2010 Dec;1(4):328-33. doi: 10.1007/s13193-011-0067-5. Epub 2011 Apr 2. PMID 22693384
- [Background] Murray JD, Elwood ET, Jones GE, Barrick R, Feng J. Decreasing expander breast infection: A new drain care protocol. Can J Plast Surg. 2009 Spring;17(1):17-21. PMID 20190908
- [Background] Carcoforo P, Soliani G, Maestroni U, Donini A, Inderbitzin D, Hui TT, Lefor A, Avital I, Navarra G. Octreotide in the treatment of lymphorrhea after axillary node dissection: a prospective randomized controlled trial. J Am Coll Surg. 2003 Mar;196(3):365-9. doi: 10.1016/S1072-7515(02)01757-X. PMID 12648685
- [Background] Park JE, Nigam M, Shenaq DS, Song DH. A simple, safe technique for thorough seroma evacuation in the outpatient setting. Plast Reconstr Surg Glob Open. 2014 Oct 7;2(9):e212. doi: 10.1097/GOX.0000000000000179. eCollection 2014 Sep. PMID 25426395
- [Background] Puttawibul P, Sangthong B, Maipang T, Sampao S, Uttamakul P, Apakupakul N. Mastectomy without drain at pectoral area: a randomized controlled trial. J Med Assoc Thai. 2003 Apr;86(4):325-31. PMID 12757076
- [Background] Rose JF, Zafar SN, Ellsworth Iv WA. Does Acellular Dermal Matrix Thickness Affect Complication Rate in Tissue Expander Based Breast Reconstruction? Plast Surg Int. 2016;2016:2867097. doi: 10.1155/2016/2867097. Epub 2016 Apr 12. PMID 27190645
- [Background] Zeidler KR, Capizzi PJ, Pittman TA. Sientra AlloX2 Short-Term Case Study, Surgical Pearls, and Roundtable Discussion. Plast Reconstr Surg. 2018 Apr;141(4S Sientra Shaped and Round Cohesive Gel Implants):29S-39S. doi: 10.1097/PRS.0000000000004352. PMID 29595716
- [Background] Moyer KE, Potochny JD. Technique for seroma drainage in implant-based breast reconstruction. J Plast Reconstr Aesthet Surg. 2012 Dec;65(12):1614-7. doi: 10.1016/j.bjps.2012.06.016. Epub 2012 Jul 6. PMID 22770571
- [Background] Jordan SW, Khavanin N, Kim JYS. Seroma in Prosthetic Breast Reconstruction. Plast Reconstr Surg. 2016 Apr;137(4):1104-1116. doi: 10.1097/01.prs.0000481102.24444.72. PMID 27018665